CLINICAL TRIAL: NCT02015000
Title: Surgical Result of Primary/Recurrent Pterygium by Pterygium Extended Removal Followed by Fibrin Glue Assisted Amniotic Membrane Transplantation
Brief Title: Surgical Result of Pterygium Extended Removal Followed by Fibrin Glue Assisted Amniotic Membrane Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201306012RINC
Record Dates: First submitted 2013-12-08; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Pterygium; Recurrence
Keywords: Pterygium; Recurrence
MeSH Terms: conditions — Pterygium; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pterygium recurrence (Experimental): Surgical Result of Primary and Recurrent Pterygium by Using Pterygium Extended Removal followed by Fibrin Glue Assisted Amniotic Membrane Transplantation (P.E.R.F.A.M.T)
  Interventions: Procedure: P.E.R.F.A.M.T

INTERVENTIONS:
Procedure: P.E.R.F.A.M.T — Surgical Result of Primary and Recurrent Pterygium by Using Pterygium Extended Removal followed by Fibrin Glue Assisted Amniotic Membrane Transplantation (P.E.R.F.A.M.T)

SUMMARY:
The treatment of pterygium is still quite controversial. Previous studies using a large incision for pterygium excision and a large graft and has reported a very low recurrence rate with the P.E.R.F.E.C.T. technique. However, the P.E.R.F.E.C.T. technique is a relatively lengthy procedure and may not be suitable for patient with limited conjunctival reserve. Thus, we try to evaluate the final outcome of a sutureless amniotic membrane transplant technique combining the extended pterygium excision in hope to avoid the complication of the P.E.R.F.E.C.T. for PTERYGIUM technique.

DETAILED DESCRIPTION:
The treatment of pterygium is still quite controversial. There is a lack of consensus in the ophthalmological community about the optimal surgical management of pterygia. The main challenge to successful surgical treatment of pterygium is recurrence, evidenced by fibrovascular growth across the limbus onto the cornea.

Previous studies using a large incision for pterygium excision and a large graft and has reported a very low recurrence rate with the P.E.R.F.E.C.T. technique. However, the P.E.R.F.E.C.T. for PTERYGIUM technique is not that perfect since it is a lengthy procedure, requires meticulous handling of tissue, and is associated with significant postoperative pain and, frequently, transient diplopia. Therefore, we try to evaluate the final outcome of a sutureless amniotic membrane transplant technique combining the extended pterygium excision in hope to avoid the complication of the P.E.R.F.E.C.T. for PTERYGIUM technique. This sutureless technique with the tissue glue may promote increased clinical use of amniotic membrane patch by alleviating patients' pain and shortening surgical time.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pterygium
* Operated by single surgeon (Chen, Wei-Li)

Exclusion Criteria:

* Follow-up time less than 12 months
* Age less then 18 year-old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pterygium | 1 year
  defined as proliferating conjunctival tissue was found extending the limbus more than 1 mm onto the cornea within the surgical field )

SECONDARY OUTCOMES:
caruncular morphology | 1 year
  A grading scale of 1 to 4 for the caruncle morphological characteristics was designed. Grade 1 with a normal appearance of the operated site; Grade 2 with the presence of fine episcleral vessels in the excised area, extending to the limbus, but without any fibrous tissue; Grade 3 with fibrovascular tissue in the excised area, reaching to the limbus but not invading the cornea; Grade 4 with aA true corneal recurrence, with fibrovascular tissue invading the cornea and across the limbus.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei City, Taiwan

REFERENCES:
- [Background] Hirst LW. Prospective study of primary pterygium surgery using pterygium extended removal followed by extended conjunctival transplantation. Ophthalmology. 2008 Oct;115(10):1663-72. doi: 10.1016/j.ophtha.2008.03.012. Epub 2008 Jun 16. PMID 18555531
- [Background] Hirst LW. Recurrent pterygium surgery using pterygium extended removal followed by extended conjunctival transplant: recurrence rate and cosmesis. Ophthalmology. 2009 Jul;116(7):1278-86. doi: 10.1016/j.ophtha.2009.01.044. PMID 19576496